CLINICAL TRIAL: NCT07156877
Title: IsoLation of PuLmonary Vein oUtcome Using a coMbIned Pulse Field Energy and ballooN cAtheTEr in Atrial Fibrillation
Brief Title: Assessment of Pulmonary Vein Isolation Using a Balloon Catheter With Pulsed Field Energy in Atrial Fibrillation
Acronym: ILLUMINATE-AF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sebastien Knecht (Other)
Responsible Party: Sponsor-Investigator, Sebastien Knecht, Coordinating investigator, AZ Sint-Jan AV
Organization: AZ Sint-Jan AV (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILLUMINATE-AF
Record Dates: First submitted 2025-08-07; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Atrial Fibrillation (AF)
Keywords: Atrial fibrillation; Pulmonary vein isolation; Pulsed field ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Desmoglein 1; Cryosurgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulsed Field Ablation (PFA) Arm - VOLT Catheter (Experimental): Participants randomized to this group will undergo pulmonary vein isolation using the novel VOLT catheter, which delivers non-thermal pulsed field energy to ablate heart tissue. The VOLT catheter features a balloon-in-basket design and is compatible with electro-anatomical mapping systems. This technique aims to selectively target heart tissue while minimizing damage to surrounding structures.
  Interventions: Procedure: Pulsed Field Ablation (PFA) with VOLT Catheter
- Thermal Ablation Arm - Radiofrequency or Cryoablation (Active Comparator): Participants in this group will receive conventional thermal ablation, either using radiofrequency energy (point-by-point ablation guided by mapping) or cryoballoon ablation (freezing tissue using a balloon catheter). These techniques create scar tissue to block abnormal electrical signals causing atrial fibrillation.
  Interventions: Procedure: Thermal Ablation (Radiofrequency or Cryoablation)

INTERVENTIONS:
Procedure: Pulsed Field Ablation (PFA) with VOLT Catheter — Participants in this arm will undergo pulmonary vein isolation (PVI) using the VOLT catheter, a novel single-shot ablation device that delivers pulsed field energy (a non-thermal ablation method). The catheter features a balloon-in-basket design and enables electro-anatomical mapping. The procedure is performed under conscious sedation or general anesthesia and follows standard PVI protocols adapted for the PFA technology.
  Arms: Pulsed Field Ablation (PFA) Arm - VOLT Catheter
Procedure: Thermal Ablation (Radiofrequency or Cryoablation) — Participants in this arm will receive PVI using established thermal ablation techniques, either:
  * Radiofrequency ablation, a point-by-point technique using heat delivered through a catheter tip guided by mapping systems, or
  * Cryoballoon ablation, which uses freezing energy delivered via a balloon catheter.
  The choice between RF and cryoablation is at the discretion of the treating physician, in line with standard care.
  Arms: Thermal Ablation Arm - Radiofrequency or Cryoablation

SUMMARY:
The goal of this clinical trial is to evaluate whether pulsed field ablation (PFA) using the novel VOLT catheter is as safe and effective as conventional thermal ablation (radiofrequency or cryotherapy) for the treatment of atrial fibrillation (AF) in adult patients undergoing their first pulmonary vein isolation (PVI).

The main questions it aims to answer are:

* Is PFA with the VOLT catheter non-inferior to thermal ablation in preventing recurrence of atrial tachyarrhythmias 2-12 months after the procedure?
* Is PFA with the VOLT catheter associated with fewer or comparable serious complications (such as cardiac tamponade, stroke, or phrenic nerve injury)?

Researchers will compare the outcomes between patients receiving PFA with the VOLT catheter and those treated with thermal ablation techniques to see if PFA offers comparable or potentially better safety and efficacy.

Participants will:

* Be randomly assigned (1:1) to receive either pulsed field ablation (PFA) or thermal ablation (radiofrequency or cryotherapy).
* Undergo standard follow-up visits at 2-3 months, 6 months, and 12 months post-ablation.
* Have repeated ECGs and Holter monitoring to assess heart rhythm.
* Complete quality of life questionnaires at baseline, 3, 6, and 12 months.
* Use a home ECG device (Kardia Mobile) weekly during the final 3 months of the study.

The study includes 136 adults (≥18 years) with paroxysmal or persistent AF, in two participating hospitals. The total study duration is 3 years, including a 2-year enrollment period and 1-year follow-up per participant.

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal or persistent atrial fibrillation documented on a 12 lead electrocardiogram or Holter monitor (lasting ≥30 seconds) within the last 24 months.
* Candidate for ablation based on current AF guidelines
* Continuous anticoagulation with Vitamin-K-Antagonists or a non-vitamin K antagonist anticoagulant (NOAC) for ≥4 weeks prior to the ablation; or a transesophageal echocardiogram (TEE) and/or computed tomography (CT) that excludes left atrial thrombus ≤48 hours before ablation
* Age of 18 years or older on the date of consent
* Informed consent as documented by signature

Exclusion Criteria:

* History of left atrial (LA) ablation or surgery involving the LA
* Persistent atrial fibrillation (AF) lasting longer than 12 months
* AF resulting from temporary or reversible causes
* Presence of thrombus within the heart chambers
* Prior pulmonary vein (PV) stenosis or stenting
* Existing paralysis of one side of the diaphragm
* Known allergy or contraindication to anticoagulant medication or contrast agents
* History of mitral valve surgery
* Significant mitral valve disease
* Myocardial infarction occurring within three months prior to informed consent
* Current use of triple antithrombotic therapy
* Cardiac surgery within the past three months or a scheduled cardiac surgery or TAVI
* Major congenital heart abnormalities
* Congestive heart failure classified as NYHA class III or IV
* Left ventricular ejection fraction (LVEF) less than 35%
* Diagnosed hypertrophic cardiomyopathy (wall thickness exceeding 1.7 cm)
* Severe chronic kidney disease (eGFR below 30 ml/min)
* Uncontrolled hyperthyroidism
* Stroke or transient ischemic attack (TIA) within three months before consent
* Active systemic infections
* History of cryoglobulinemia
* Diagnosed cardiac amyloidosis
* Current pregnancy
* Estimated life expectancy under one year, as judged by the treating physician
* Enrollment in another clinical study that may interfere with this trial's outcomes
* Inability or unwillingness to adhere to study requirements and follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Time to first recurrence of any atrial tachyarrhythmia | Between 2 and 12 months post ablation
  The primary endpoint is the time to first recurrence of any atrial tachyarrhythmia (AF and/or organized atrial tachyarrhythmia) after 12 months following the ablation procedure, as detected on repetitive Holter and home monitoring. During the first 2 months after the procedure (blanking period), recurrent AF or atrial tachycardia will be treated with antiarrhythmic drugs or cardioversion as needed, and won't be considered treatment failure.
  Atrial tachyarrhythmia recurrence is defined as continuous arrhythmia lasting 30 seconds or longer. Potential arrhythmia events will be independently reviewed and adjudicated by a clinical events committee comprised of 3 experienced electrophysiologists who are blinded to treatment allocation.
Number of safety events, composite of cardiac tamponade, phrenic nerve palsy, vascular complications, stroke/transient ischemic attack, atrio-esophageal fistula and death | From ablation until 30 days post ablation
  The primary safety endpoint is a composite of:
  1. Cardiac tamponade requiring pericardiocentesis
  2. Persistent phrenic nerve palsy lasting more than 24 hours
  3. Serious vascular complications requiring intervention
  4. Stroke/transient ischemic attack
  5. Atrio-esophageal fistula
  6. Death The safety endpoint is assessed during catheter ablation, until discharge, and during the following 30 days. Information on safety events are collected throughout the trial by the investigators or their designees. All primary safety events will be reviewed and adjudicated by the clinical events committee members.
Procedure duration (minutes) | Day of ablation procedure
  Total procedure duration (minutes)

SECONDARY OUTCOMES:
Left atrial dwelling time (minutes) | Day of ablation procedure
  Time the catheter remains inside the left atrium during the ablation procedure (minutes)
Fluoroscopy time (minutes) | Day of ablation procedure
  Total fluoroscopy time (minutes)
AF burden: percentage of time in AF on 7 day Holter (%) | Before ablation, and 6 months and 12 months post ablation
  AF burden: percentage of time in AF on 7 day Holter (%)
Proportion of patients with recurrence of any atrial tachyarrhythmia including during the blanking period (%) | From ablation until 12 months post ablation
  Proportion of patients with recurrence of any atrial tachyarrhythmia including during the blanking period (%)
Proportion of patients undergoing a repeat ablation (%) | From ablation until 12 months post ablation
  Proportion of patients undergoing a repeat ablation (%)
Quality of life changes, assessed using the 36-Item Short Form Survey Instrument (SF-36) | 3, 6 and 12 months post ablation
  Quality of life changes at 3, 6 and 12 months compared with baseline, assessed using the 36-Item Short Form Survey Instrument (SF-36)
Quality of life changes, assessed using the AF Symptom Checklist | 3, 6 and 12 months post ablation
  Quality of life changes at 3, 6 and 12 months compared with baseline, assessed using the AF Symptom Checklist

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Knecht, MD, PhD, Principal Investigator — AZ Sint-Jan Brugge AV
Locations (2):
- Belgium (2):
  - AZ Sint-Jan Brugge AV, Bruges
  - UZ Brussel, Jette

IPD SHARING:
Plan to Share IPD: No